CLINICAL TRIAL: NCT00582400
Title: A Phase II Protocol of Arsenic Trioxide (Trisenox) in Subjects With Advanced Primary Carcinoma of the Liver
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruiting or enrolling participants has halted prematurely and will not resume; participants are no longer being examined or treated
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-267; PI-Initiated
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2010-01

CONDITIONS: Carcinoma, Hepatocellular
Keywords: livers, hepatocellular carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental)
  Interventions: Drug: arsenic trioxide

INTERVENTIONS:
Drug: arsenic trioxide — Trisenox will be diluted with 100 to 250 mL 0.9% Sodium Chloride injection, USP, using proper aseptic technique, immediately after withdrawal from the ampule. The Trisenox ampule is single-use and does not contain any preservatives. Unused portions of each ampule should be discarded properly. Trisenox is not to be mixed with other medications.
  The loading dose of Trisenox will be administered intravenously over 2 hours. The infusion duration may be extended up to 4 hours if acute vasomotor reactions are observed. The drug will be administered IV through a functional peripheral or central venous line. Trisenox is not a vesicant, and may be a mild irritant if administered into the skin without dilution.
  Other Names: Trisenox

SUMMARY:
The purpose of this study is: evaluate the safety and activity of administering arsenic trioxide (Trisenox) in the treatment of unresectable or metastatic primary liver cancer, to evaluate the qualitative and quantitative toxicities of this treatment, and to measure the response to treatment and the patterns of failure and survival. The primary response measurements will be the achievement of an objective tumor response, response duration and progression-free survival

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most frequently diagnosed malignancies in some regions of the world, particularly Africa and the Asian portion of the Pacific rim. However, it is an uncommon malignancy in the United States, with less than 14,000 cases diagnosed annually. Malignancies of the gallbladder and biliary tree are also uncommon. As with most solid tumors, unless either neoplasm can be resected completely, the prognosis is grim. A variety of agents have been utilized in the therapy of HCC and cholangiocarcinoma, both as single agents and in combination regimens. However, despite response rates which exceed 50% when hepatic arterial therapy is utilized for HCC, response rates for cholangiocarcinoma and for systemic treatment of HCC are considerably lower. Long term survival remains uncommon. For this reason, new therapeutic approaches must be evaluated.

Trisenox (arsenic trioxide) is a newly-approved pharmaceutical grade arsenic compound antineoplastic agent which has demonstrated clear activity in anthracycline- and all-trans retinoic acid-resistant acute promyelocytic leukemia. Trisenox also has US Compendium listing for acute leukemia, chronic myelogenous and lymphocytic leukemias, myelodysplasia, multiple myeloma, and hepatocellular carcinoma (HCC). Similar to the taxanes and vinca alkaloids, Trisenox appears to interfere with microtubule function, which triggers cell differentiation, and induces programmed death, or apoptosis. The mechanism of this is unclear, but appears to involve activation of caspases and the down-regulation of the BCL-2 oncogene. Trisenox also interfere with the function of NF-kappaB, leading to inhibition of cellular proliferative signals, apoptosis, and inhibition of tumor angiogenesis.

Trisenox was shown to be effective in a pivotal trial consisting of 40 subjects, ages 5 to 72, at a nine-institution multi-center trial led by Memorial Sloan-Kettering Cancer Center. With Trisenox, 70% of the subjects achieved a complete remission, and 79% of the complete responders achieved a molecular remission as measured by reverse transcriptase-polymerase chain reaction (RT-PCR). Complete remission was achieved on average within two months after initiation of Trisenox. Sixty-eight percent of subjects who achieved complete remission were still alive and 58% were disease free, at a median follow-up time of 16 months.

To date, an optimal dose and schedule of Trisenox has not yet been defined. This agent has been administered on daily, twice a week, and weekly doses. As there is no evidence that one regimen is clearly superior to any other, for the sake of convenience, participants on this trial will receive Trisenox on the weekly schedule. Administration of chemotherapy on a weekly schedule is commonly utilized across a broad spectrum of regimens and tumor types. On this trial, subjects will receive a dose of intravenous Trisenox 0.35 mg/kg on days 1, 8, 15, and 22 over two hours. Each cycle will be 28 days in length. Subjects will receive two treatment cycles (8 weeks) and then undergo objective radiographic tumor assessments. On this study, subjects may receive up to a maximum of 12 such treatment cycles. As the outlook for subjects with advanced primary liver cancer is so poor, new regimens and treatment strategies must be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* ECOG/Zubrod/SWOG Performance Status < 2
* Life expectancy > 12 weeks
* Male or female' age >18 years Subjects of childbearing potential must be using an effective means of contraception.
* Histologic diagnosis of HCC or cholangiocarcinoma that is locally advanced but cannot be treated adequately by radiotherapy or surgery (more than one lesion, portal vein involvement, or poor hepatic reserve); or metastatic disease or an AFB > 20 w/CT scan consistent with HCC
* Renal function: Serum creatinine < 2.0 mg/dl
* Serum calcium < 12 mg/dl
* Serum electrolytes, including magnesium and potassium, within normal limits

Exclusion Criteria:

* Pregnant or lactating females
* Myocardial infarction or ischemia within the 6 months before Cycle 0' Day 0
* Uncontrolled' clinically significant dysrhythmia
* Known left ventricular Ejection Fraction below the normal limit for UTMB
* History of prior malignancy within the prior five years, with the exception of non-melanoma carcinomas of the skin, and carcinoma in situ of the cervix
* More than one prior chemotherapy regimens for liver cancer (subjects who are receiving antineoplastic agents for non-malignant conditions, such as methotrexate for rheumatoid arthritis, must be off such therapy for at least four weeks prior to receiving the first dose of protocol therapy, and may not receive such therapy while participating in this protocol)
* Receiving any other chemotherapy or cytokine therapy
* Subjects receiving radiation therapy (Trisenox will be held during the administration of palliative or emergent radiotherapy)
* Subjects who have received radiofrequency ablation or hepatic arterial embolization within the past four weeks (patients who have received prior RFA or HAE are otherwise eligible)
* Prior radiotherapy to an indicator lesion unless there is objective evidence of tumor growth in that lesion
* Uncontrolled metastatic disease of the central nervous system
* Prior and on-going Grade 2-4 peripheral neuropathy, as measured by NCI Common Toxicity Criteria version 3.0
* Radiotherapy within the 2 weeks before Cycle 1' Day 1
* Surgery within the 2 weeks before Cycle 1' Day 1
* Any co morbid condition that' in the view of the attending physician' renders the subject at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avi B. Markowitz, MD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch at Galveston, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine patients were enrolled from 10/13/04 to 09/05/07 from the outpatient clinics (both free-world and prisoners). The median age of patients was 57 years (range 50-62) and included 8 males and 1 female.
Pre-assignment Details: No patients had previous systemic therapy.
Groups:
- Arsenic Trioxide: Patients with advanced measurable HCC, no more than one prior systemic treatment or no treatment, ECOG PS 0-2, and Child-Pugh class A received arsenic trioxide 0.35mg/kg on days 1, 8, 15 and 22 of each 28-day cycle.
Period: Overall Study
Arm/Group | Arsenic Trioxide
Started | 9
Completed | 6
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 57 [50 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Toxicity.
Time Frame: 6 years
Measure: Number; unit: participants
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 9
participants | 0

2. Primary Outcome: Number of Patients With Response to Treatment (RECIST Criteria)
Description: Response included complete response, partial response or stable disease.
Time Frame: 6 years
Population: Participants who were evaluable for response
Measure: Number; unit: participants
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 7
participants | 1

3. Secondary Outcome: Duration of Response.
Description: Time to progression.
Time Frame: 6 years
Population: Participants with response
Measure: Median (Full Range); unit: months
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 1
months | 8 [8 to 8]

4. Secondary Outcome: Progression Free Survival
Description: Time to progression from start of treatment
Time Frame: 6 years
Population: 1 evaluable participant lost to follow up. No data collected.
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Arsenic Trioxide (Trisenox): arsenic trioxide: Trisenox will be diluted with 100 to 250 mL 0.9% Sodium Chloride injection, USP, using proper aseptic technique, immediately after withdrawal from the ampule. The Trisenox ampule is single-use and does not contain any preservatives. Unused portions of each ampule should be discarded properly. Trisenox is not to be mixed with other medications.
  The loading dose of Trisenox will be administered intravenously over 2 hours. The infusion duration may be extended up to 4 hours if acute vasomotor reactions are observed. The drug will be administered IV through a functional peripheral or central venous line. Trisenox is not a vesicant, and may be a mild irritant if administered into the skin without dilution.
Arm/Group | Arsenic Trioxide (Trisenox)
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arsenic Trioxide (Trisenox) (N=9)
hemorrhagic diarrhea (Gastrointestinal disorders) | 1 (1) — Blood in stool
abdominal pain (Gastrointestinal disorders) | 1
bilateral extremity edema (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arsenic Trioxide (Trisenox) (N=9)
abdominal pain (Gastrointestinal disorders) | 1 (1) — abdominal pain and swelling
abdominal edema (Gastrointestinal disorders) | 1 (1)
bilateral lower extremity weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No